CLINICAL TRIAL: NCT03771144
Title: Anatomopathology of the Subscapularis and Infraspinatus Muscles in Children With Brachial Plexus Obstetric Paralysis
Acronym: POPB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator's decision
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL18_0175
Record Dates: First submitted 2018-11-30; First posted 2018-12-10 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Brachial Obstetrical Palsy
Keywords: Brachial obstetrical palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Procedure: arthrolysis

INTERVENTIONS:
Procedure: arthrolysis — Surgery is performed under general anesthesia. The usual duration of this surgery is on average 1h30. This surgery requires an anterior approach and a posterior approach. The patient is placed in lateral decubitus. The arthroscope of 2.7 is introduced by a posterior route. An anterior instrumental track is made from inside out through the rotator interval.

SUMMARY:
POPB is a consequence of the stretching of the nerve roots (C5, C6 + / C7, C8 or T1) of the brachial plexus at birth. One third of patients will have sequelae. The most common is the appearance of a deficit of passive and active mobilities in the movements in external rotation of the shoulder especially in external rotation (RE) elbow to the body, despite daily rehabilitation. At present, this stiffness is attributed to an imbalance between the external rotator muscles (mainly infraspinatus) that would be atrophied and the internal rotator muscles (subscapularis, pectoralis major, latissimus dorsi) that would be slightly affected In case of no or negative RE from the age of 1 year, there is a surgical indication to operate these children. At present, surgery to lift internal retractions is the only therapy used, but despite this surgery and intensive rehabilitation, in some patients mobility deficits re-occur in a few years. Thus, some teams systematically perform a muscle transfer to strengthen the outer rotator muscles deficit during the initial operation. Other teams (of which principal investigator is part) do this transfer only secondarily and in some patients. Investigators lack objective and scientific criteria for the indication of this second muscle transfer surgery and the etiology of retractions is not clearly defined.

In humans, subscapularis is innervated by the C5 and C6 roots, which are constantly affected in POPB. It can be assumed that subscapularis may have an atrophy in POPB patients. To date, no anatomopathological study has been performed on the internal / external rotator muscles of patients with POPB that can give indications on recurrences.

Based on our clinical observations and literature data, the main hypothese is there is amyotrophy of subscapularis and / or infraspinatus in POPB patients with shoulder stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Child with POPB presenting a stiffness in external shoulder rotation after the age of 1 year with a surgical indication of anterior release of shoulder is asked
* Obligation to obtain written informed consent from parents.

Exclusion Criteria:

* Patient with another neuromuscular pathology
* Significant traumatic history of the upper limb (fracture or surgical intervention) or any other pathology affecting the mobility of the joints of the upper limb (either on the pathological side or on the healthy side)
* Patient with a contraindication to surgery (precarious general condition, major coagulation disorders, anesthetic contraindication)
* Child over 10 years old
* Refusal of the patient or family

Ages: 12 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
quantity of fibrosis on tissue muscle | 1 day

SECONDARY OUTCOMES:
quantity of satellit cells (Pax7, MyoD,Actine) on the muscle detected by PCR | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No